CLINICAL TRIAL: NCT01558492
Title: A Phase II Trial of Carboplatin and Paclitaxel in Patients With Metastatic, Castrate-Resistant Prostate Cancer Previously Treated With Docetaxel
Brief Title: Carboplatin and Paclitaxel in Patients With Metastatic, Castrate-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008011188
Record Dates: First submitted 2012-02-16; First posted 2012-03-20 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: Metastatic Castrate Resistant Prostate Cancer; CRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental): Carboplatin and Paclitaxel
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — AUC = 5 intravenously (IV) on day 1 of a 28 day cycle
  Other Names: Paraplatin
Drug: Paclitaxel — 80 mg/m2 intravenously (IV) weekly on days 1, 8, and 15 of a 28 day cycle
  Other Names: Taxol

SUMMARY:
The purpose of this study is to look at the clinical benefit of carboplatin and paclitaxel and correlate response to study treatment with biologic parameters (i.e. lab studies of blood, urine, or tissue). It is hoped that this will allow researchers to gain insight into the underlying biology of prostate tumor progression and perhaps predict which patients may benefit from this chemotherapy regimen.

DETAILED DESCRIPTION:
Docetaxel/prednisone is the standard of care in patients with metastatic, castrate-resistant prostate cancer (CRPC) but duration of response is limited, with median time to prostate-specific antigen (PSA) progression of 6-8 months. There is currently no standard second-line therapy for patients who have progressed after receiving docetaxel. Carboplatin and paclitaxel have demonstrated activity, but prospective clinical trials evaluating this regimen are limited. In addition, correlative studies investigating why some patients respond are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of prostate carcinoma.
* Subject must have progressive metastatic prostate cancer despite adequate medical or surgical castration therapy. Furthermore, if applicable, medical castration must be maintained for the duration of the protocol.
* Serum testosterone < 50 ng/ml.
* Subjects who have received anti-androgen therapy with a resulting PSA decline must demonstrate progression following discontinuation of anti-androgen therapy.
* Subjects capable of fathering children must agree to use an effective method of contraception for the duration of the trial.
* Must have previously received docetaxel for prostate cancer
* ECOG performance status 0-2
* Willing and able to give informed consent

Exclusion Criteria:

* Platelet count <100,000/mm3
* Absolute neutrophil count (ANC) <1,500/mm3
* Hemoglobin < 8 g/dL
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x upper limit of normal
* Bilirubin (total) >2 x upper limit of normal. Subjects with known Gilbert's syndrome are eligible if direct bilirubin is within normal limits
* For subjects with serum creatinine > 1.5 x ULN, calculated creatinine clearance < 30 ml/min are excluded; subjects meeting this exclusion criterion are eligible if a measured clearance is > 30 ml/min
* Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
* Prior investigational therapy within 4 weeks of treatment. Furthermore, other investigational anti-cancer therapy is not permitted during the treatment phase.
* Grade > 1 peripheral neuropathy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himisha Beltran, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Prostate-specific Antigen (PSA) Level
Time Frame: Baseline, week 4, week 8, week 12, week 16, week 20, week 24 and end of study.
Population: This study was terminated early due to poor accrual. There were no publications as a result. Data were not collected.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Tumor Size
Description: Assessed by CT or MRI scan and/or bone scan.
Time Frame: Baseline, week 12, week 24 and end of study.
Population: This study was terminated early due to poor accrual. There were no publications as a result. Data were not collected.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Survival Status
Time Frame: 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months and 48 months.
Population: This study was terminated early due to poor accrual. There were no publications as a result. Data were not collected.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes